CLINICAL TRIAL: NCT03010462
Title: A Prospective, Multi-center, Randomized, Sham-controlled Trial to Determine the Therapeutic Effects of Navigation Guided 1 hz Rtms Administered to the Contralesional Hemisphere as Adjuvant to Task-oriented Rehabilitation in Patients With Ischemic Stroke
Brief Title: Electric Field Navigated 1hz Rtms for Post-stroke Motor Recovery Trial
Acronym: E-FIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nexstim Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NX103391
Record Dates: First submitted 2017-01-03; First posted 2017-01-05 (Estimated); Results first posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-03

CONDITIONS: Ischemic Stroke
Keywords: Stroke; rTMS; Motor rehabilitation
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active (Active Comparator): Intervention: Device: NBS-guided rTMS + task-oriented rehabilitation
  Interventions: Device: Nexstim NBS guided active rTMS
- Control (Sham Comparator): Intervention: Device: NBS-guided Sham rTMS + task-oriented rehabilitation
  Interventions: Device: Nexstim NBS guided sham rTMS

INTERVENTIONS:
Device: Nexstim NBS guided active rTMS — Nexstim NBS guided active rTMS + standardized task-oriented therapy
  Arms: Active
Device: Nexstim NBS guided sham rTMS — Nexstim NBS guided sham rTMS + standardized task-oriented therapy
  Arms: Control

SUMMARY:
A prospective, multi-center, randomized, sham-controlled, blinded study combining active Nexstim NBS-guided 1Hz rTMS or sham-rTMS targeting the healthy hemisphere with standardized task oriented rehabilitation will be conducted in patients with post-stroke motor impairment of the upper limb. The therapy will be provided for 6 weeks and primary outcome assessed 6 months later.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* An ischemic stroke suffered 3-12 months prior to the study
* No other known brain abnormalities by history;
* A one-sided stroke resulting in upper extremity paresis
* A Chedoke-McMaster Stroke Assessment arm stage and hand stage of 3-6 for the affected limb

Exclusion Criteria:

* Implanted metallic parts of implanted electronic devices, including pacemakers, defibrillators, or implant medication pump;
* Pregnant or trying to become pregnant; Lack of pregnancy established in females of child-bearing potential by a negative urine pregnancy test at screening.
* Active alcohol abuse, illicit drug use or drug abuse or significant mental illness
* Patients suffering from depression as measured by a score of >10 on the Patient Health Questionnaire (PHQ9). For clarity, patients diagnosed with depression which is controlled with stable anti-depressive medication and in whom PHQ9 is <10 are eligible to participate in the trial.
* History of epilepsy, defined as at least two unprovoked seizures occurring greater than 24 hours apart or diagnosis of an epilepsy syndrome, OR a seizure within the last 12 months.
* Any condition that would prevent the subject from giving voluntary informed consent;
* An implanted brain stimulator;
* Any metal in head with the exception of dental work or any ferromagnetic metal -elsewhere in the body;
* Enrolled or plans to enroll in an interventional trial during this study;
* Scalp wounds or infections;

  * Claustrophobia precluding MRI;
* A fixed contraction deformity in the affected limb that would prevent normal dexterity if patient were neurologically intact;
* Excessive spasticity as indicated by the Modified Ashworth Spasticity (MAS) Scale >2/4 in either elbow flexors, wrist flexors or finger flexors of the affected limb;
* Previous stroke with residual deficits (TIAs not a reason for exclusion);
* Premorbid (retrospective) modified Rankin Scale (mRS) score ≥2 of any aetiology;
* A concurrent progressive neurologic disorder, acute coronary syndrome, severe heart disease (NYHA Classification > 3), or other major medical condition,
* Confirmed or suspected lower-limb fracture preventing mobilization, patients requiring palliative care
* Patients planning to undergo any other occupational therapy during the 6 week active treatment period of the trial (see section 5.2 for study schedule) than what is provided in the study
* A recent injection of botulinium toxin to the affected upper limb in the last 3 months, or the need of an injection of botulinum toxin anytime during the study period and follow up.
* A recent injection of phenol to the affected upper limb in the last 6 months, or the need of an injection of phenol anytime during the study period and follow up.
* Ataxia as measured by a score > 1 on item 7 (limb ataxia) of the NIH stroke scale.
* Severe sensory deficits as measured by a score of 2 on item 8 of the NIH stroke scale.
* Severe aphasia as measured by a score of > 2 on item 9 (best language) of the NIH stroke scale.
* Severe neglect as measured by a score of 2 on item 11 (extinction and inattention) of the NIH stroke scale.
* Patients unable to comprehend or follow verbal commands
* Based on PI's or local physician's assessment patient unable to tolerate the trial procedure due to medical condition
* A Mini mental status exam (MMSE) <25.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Rancho Los Amigos National Rehabilitation Center, Downey, California
  - Rehabilitation Institute of Chicago, Chicago, Illinois
  - Spaulding Rehabilitation Hospital, Boston, Massachusetts
  - Burke Medical Research Institute, Weill Cornell Neurology, White Plains, New York
  - University of Cincinnati, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Edwards DJ, Liu CY, Dunning K, Fregni F, Laine J, Leiby BE, Rogers LM, Harvey RL. Electric Field Navigated 1-Hz rTMS for Poststroke Motor Recovery: The E-FIT Randomized Controlled Trial. Stroke. 2023 Sep;54(9):2254-2264. doi: 10.1161/STROKEAHA.123.043164. Epub 2023 Aug 14. PMID 37577801

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active | Control
Started | 31 | 29
Completed | 28 (1 subject withdrew consent before baseline visit. 2 subjects completed treatment but were lost during follow-up) | 28 (1 subject withdrew consent prior to baseline visit)
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Control | Total
Number analyzed (Participants) | 31 | 29 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (9.5) | 58.0 (10.9) | 58.5 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 23 | 19 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 9 | 15
  White | 24 | 20 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Time from stroke [Count of Participants; unit: Participants]
  3-6 months | 15 | 12 | 27
  6-12 months | 16 | 17 | 33
Upper extremity Fugl-Meyer score [Mean (Standard Deviation); unit: units on a scale] — Population: 2 subjects ( 1 active, 1 sham withdraw consent prior to analysis of study specific baseline characteristics)
  units on a scale
    number analyzed (Participants) | 30 | 28 | 58
    (all) | 37.4 (12.7) | 42.2 (13.2) | 39.7 (13.1)
Action Research Arm Test [Mean (Standard Deviation); unit: units on a scale] — Population: 2 subjects ( 1 active, 1 sham withdraw consent prior to analysis of study specific baseline characteristics)
  units on a scale
    number analyzed (Participants) | 30 | 28 | 58
    (all) | 28.9 (17.7) | 34.7 (16.7) | 31.7 (17.3)
NIHSS [Mean (Standard Deviation); unit: units on a scale] — Population: 2 subjects ( 1 active, 1 sham withdraw consent prior to analysis of study specific baseline characteristics)
  units on a scale
    number analyzed (Participants) | 30 | 28 | 58
    (all) | 2.23 (1.74) | 1.86 (1.88) | 2.05 (1.80)
EQ-5D [Mean (Standard Deviation); unit: units on a scale] — Population: 2 subjects ( 1 active, 1 sham withdraw consent prior to analysis of study specific baseline characteristics)
  units on a scale
    number analyzed (Participants) | 30 | 28 | 58
    (all) | 61.8 (19.9) | 70.1 (18.4) | 65.8 (19.5)

OUTCOME MEASURES:

1. Primary Outcome: Upper Extremity Fugl-Meyer Score
Description: Range 0 to 65. HIgher scores indicate better function. Minimal clinically important difference = change of 5 points or more on scale. Outcome measure = proportion of patients in treatment arm gaining at least 5 points on scale between baseline and 6 months after end of treatment.
Time Frame: Change from baseline to 6 months after end of treatment.
Population: Intent to treat population. All subjects completing the baseline visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Control
Number analyzed (Participants) | 30 | 28
Participants | 18 | 14
Statistical Analysis 1: Comparison: Active vs Control; Test type: Superiority; p = 0.62, Chi-squared, Corrected

2. Secondary Outcome: Upper Extremity Fugl-Meyer Score
Description: Range 0-65. HIgher scores indicate better function.
Time Frame: Change in score from baseline to 6 months after end of treatment
Population: Intent to treat population. All enrolled subjects who completed the baseline visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active | Control
Number analyzed (Participants) | 30 | 28
units on a scale | 5.17 (8.24) | 5.00 (7.29)
Statistical Analysis 1: Comparison: Active vs Control; Test type: Superiority; p = 0.46, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Arm-Research Action Test (ARAT)
Description: Range 0 to 57. Higher scores indicate better function.
Time Frame: Change in score from baseline to 6 months after end of treatment.
Population: Intent to treat population. All subjects completing the baseline visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active | Control
Number analyzed (Participants) | 30 | 28
units on a scale | 4.93 (6.99) | 5.68 (7.96)
Statistical Analysis 1: Comparison: Active vs Control; Test type: Superiority; p = 0.54, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: NIH Stroke Scale (NIHSS)
Description: National Institute of Health Stroke Scale - Motor Arm. Range 0 to 4. Lower score indicates better function.
Time Frame: Change in score from baseline to 6 months after end of treatment
Population: Intent to treat. All subject completing the baseline visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active | Control
Number analyzed (Participants) | 30 | 28
units on a scale | -0.62 (1.35) | -0.50 (1.40)
Statistical Analysis 1: Comparison: Active vs Control; Test type: Superiority; p = 0.59, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Quality of Life Assessment: EQ-5D
Description: EuroQoL - EQ-5D score. Range 0 to 100. HIgher numbers indicate better quality of life.
Time Frame: Change in score from baseline to 6 months after end of treatment
Population: Intent to treat - all subjects completing the baseline visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active | Control
Number analyzed (Participants) | 30 | 28
units on a scale | 9.86 (21.09) | 8.96 (18.80)
Statistical Analysis 1: Comparison: Active vs Control; Test type: Superiority; p = 0.70, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: From baseline until 6 months after end of treatment.
Arm/Group | Active | Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/28
Serious Adverse Events (participants affected / at risk) | 4/30 | 5/28
Other Adverse Events (participants affected / at risk) | 5/30 | 2/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=30) | Control (N=28)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Self-injurious ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=30) | Control (N=28)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 2 (5)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Fatigue (General disorders) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/62/NCT03010462/Prot_SAP_000.pdf